CLINICAL TRIAL: NCT01854359
Title: Open Label Extension Trial of Idebenone for Primary Progressive Multiple Sclerosis
Brief Title: Idebenone for Primary Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130088; 13-I-0088
Record Dates: First submitted 2013-05-11; First posted 2013-05-15 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis; Primary Progressive Multiple Sclerosis
Keywords: Multiple Sclerosis; Extension Trial
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — idebenone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Active treatment (Other): Idebenone (150mg tablets) administered orally as five tablets, three times per day with food.
  Interventions: Drug: Idebenone

INTERVENTIONS:
Drug: Idebenone

SUMMARY:
Background:

- The Idebenone in Patients With Primary Progressive Multiple Sclerosis (IPPoMS) trial tested a new drug for multiple sclerosis. In the IPPoMS trial, participants took either idebenone or placebo. Researchers want to give idebenone to all participants for 1 year. It is still not certain whether idebenone can slow the progression of multiple sclerosis, but this study may help answer that question.

Objectives:

* To provide idebenone to all participants on the IPPoMS trial.
* To collect data on the safety and effectiveness of idebenone for primary progressive multiple sclerosis.

Eligibility:

- Individuals at least 18 years of age who have completed 3 years in the IPPoMS trial.

Design:

* The first study visit for this trial will happen on the same day as the last visit for the IPPoMS trial.
* Participants will provide a blood samples and will have a lumbar puncture. They will also receive a new supply of idebenone to take three times a day with food. They will keep a diary to report on any side effects.
* After this first treatment visit, participants will have two follow-up visits to the NIH 6 months apart. These visits may be scheduled over multiple days. Participants will provide blood and urine samples. They will also have imaging studies of the brain and spine.
* Participants will have phone calls with the study researchers to provide updates on their condition and any side effects.

DETAILED DESCRIPTION:
OBJECTIVE:

A Phase I/II clinical trial is being conducted to investigate the safety, therapeutic efficacy and mechanism of action of idebenone in primary-progressive multiple sclerosis (PP-MS) patients (IPPoMS (Protocol Number 09-N-0197). Patients who have completed the 2-year treatment period of IPPoMS, may enter into this open-label extension study (IPPoMS-E) if they are found to be eligible by the Investigator and desire treatment with idebenone despite remaining blinded as to their allocation to active treatment versus placebo during the IPPoMS trial. The aim of this open-label extension study is gather additional data on safety, efficacy and effects of idebenone on cerebrospinal fluid (CSF) biomarkers in these patients over a period of 1 year. This study will provide open-label idebenone for patients with PP-MS, previously randomized to idebenone or to placebo in the blinded phase of IPPoMS.

STUDY POPULATION:

Patients who were previously enrolled in the IPPoMS (Protocol Number 09-N-0197) will be invited to participate in the trial. The same idebenone dose used in the randomized clinical trial (2250 mg/day) will be used in this study.

DESIGN:

This is a single group, open-label safety and efficacy extension trial with a one year treatment period. Patient-specific biomarkers of disease progression, CSF biomarkers of oxidative stress, longitudinal neuroimaging including quantitative measures of CNS tissue destruction and clinical data will be collected as in the randomized study.

OUTCOME MEASURES:

The measurement and collection of data will be performed as in the randomized trial. Quantitative neuroimaging measures of central nervous system (CNS: i.e. brain and spinal cord) tissue destruction and clinical and functional measures of neurological disability will be collected every 6-12 months. Additionally, biomarkers focusing on analysis of reactive oxygen species (ROS) and oxidative stress will be collected every 12 months. The primary outcome measure defined in the IPPoMS trial will be also utilized in IPPoMS-E. For patients originally randomized to placebo, patient-specific slopes of disease progression during 2 years of placebo therapy (as measured by primary and secondary outcomes) will be compared to patient-specific slopes of disease progression during 1 year of open label idebenone therapy. Combination of IPPoMS and IPPoMS-E trials will significantly expand paired no therapy vs. idebenone therapy CSF samples for biomarker studies. It will also provide (for the subgroup of subjects who were originally randomized to idebenone) longitudinal CSF samples on idebenone therapy (collected 2 years apart). This will allow calculations of intra-individual changes in CSF biomarkers on and off idebenone therapy, which may provide important insight into the mechanism of action of idebenone in PP-MS.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Completion of 3 years in study IPPoMS (Protocol Number 09-N-0197)
* Able to provide informed consent
* Adults, at least 18 years of age
* Willing to participate in all aspects of trial design and follow-up
* If able to become pregnant or to father a child, agreeing to commit to the use of a reliable/accepted method of birth control (i.e. hormonal contraception (birth control pills, injected hormones, vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation, or vasectomy)) for the duration of treatment arm of the study

EXCLUSION CRITERIA:

* Pregnant or lactating women. All women of child-bearing potential must have a negative pregnancy test
* Patients dropping out of IPPoMS due to adverse events (AE) considered related to study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Bielekova, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Albrecht P, Ringelstein M, Muller AK, Keser N, Dietlein T, Lappas A, Foerster A, Hartung HP, Aktas O, Methner A. Degeneration of retinal layers in multiple sclerosis subtypes quantified by optical coherence tomography. Mult Scler. 2012 Oct;18(10):1422-9. doi: 10.1177/1352458512439237. Epub 2012 Mar 2. PMID 22389411
- [Background] Andrews HE, Nichols PP, Bates D, Turnbull DM. Mitochondrial dysfunction plays a key role in progressive axonal loss in Multiple Sclerosis. Med Hypotheses. 2005;64(4):669-77. doi: 10.1016/j.mehy.2004.09.001. PMID 15694681
- [Background] Artuch R, Aracil A, Mas A, Colome C, Rissech M, Monros E, Pineda M. Friedreich's ataxia: idebenone treatment in early stage patients. Neuropediatrics. 2002 Aug;33(4):190-3. doi: 10.1055/s-2002-34494. PMID 12368988
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-I-0088.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment in 09-I-0197: Idebenone (150mg tablets) administered orally as five tablets, three times per day with food.
  This group completed a total of 3 years of Idebenone treatment
- Placebo in 09-I-0197: Idebenone (150mg tablets) administered orally as five tablets, three times per day with food.
  This group completed a total of 1 year of Idebenone treatment (following 2 years of placebo treatment in the 09-I-0198 trial).
Period: Overall Study
Arm/Group | Active Treatment in 09-I-0197 | Placebo in 09-I-0197
Started | 31 | 30
Completed | 26 | 22
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Placebo in 09-I-0197: Idebenone (150mg tablets) administered orally as five tablets, three times per day with food.
  This group completed a total of 1 year of Idebenone treatment (following 2 years of placebo treatment in the 09-I-0197 trial)
- Total: Total of all reporting groups
Arm/Group | Active Treatment in 09-I-0197 | Placebo in 09-I-0197 | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (6.7) | 59.2 (7.2) | 59.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 17 | 13 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Combinatorial Weight-Adjusted Disability Score (CombiWISE)
Description: CombiWISE is a composite scale derived from Expanded Disability Status Scale (EDSS) , Scripps Neurological Disability Scale (SNRS), times 25 foot walk (25FW), and non-dominant hand of 9 hole peg test (9HPT) with a minimum value of 0 (no disability) and maximum value of 100 (maximum disability).
  The AUC values were calculated for both study groups (Active treatment group in the 09-I-0197 trial and Placebo group in the 09-I-0197) as follows:
  1. pre-treatment baseline during the 09-I-0197 trial (from Months -12, -6, and 0)
  2. double-blind phase during the 09-I-0197 trial (from Months 0, 6, 12, 18, and 24)
  3. extension phase during the 13-I-0088 trial (from Months 24, 30, and 36)
  Because the follow-up times varied from patient to patient, the AUC values were made comparable by scaling them by dividing the AUC value by the square of the actual duration (in years) of each of the phases.
Time Frame: 1-year pre-treatment baseline vs 2-year randomized double-blind phased vs 1-year treatment period
Population: 61 subjects that completed three year 09-I-0197 trial enrolled into the one year open-label extension phase of the 13-I-0088.
  Out of the 61 subjects, 31 were assigned to the active treatment group in the 09-I-0197 trial and 30 received placebo.
  The 09-I-1097 consisted of one-year pre-treatment baseline and 2 years of double-blind treatment phase.
Measure: Mean (Standard Deviation); unit: units on a scale * year
Groups:
- Pre-treatment Baseline (Placebo Group): One Year Pre-treatment baseline of the 09-I-0197 trial for placebo group
- Double-blind Phase (Placebo Group): Two-Year Double-blind Phase of 09-I-0197 (placebo group)
- Extension Phase (Placebo Group): One-year open label active treatment group that received placebo in the 09-I-0197 trial
- Pre-treatment Baseline (Active Treatment Group): One Year Pre-treatment baseline of the 09-I-0197 trial for active treatment group
- Double-blind Phase (Active Treatment Group): Two-Year Double-blind Phase of 09-I-0197 (active treatment group)
- Extension Phase (Active Treatment Group): One-year open label active treatment group that received active treatment in the 09-I-0197 trial
Arm/Group | Pre-treatment Baseline (Placebo Group) | Double-blind Phase (Placebo Group) | Extension Phase (Placebo Group) | Pre-treatment Baseline (Active Treatment Group) | Double-blind Phase (Active Treatment Group) | Extension Phase (Active Treatment Group)
Number analyzed (Participants) | 30 | 30 | 22 | 31 | 31 | 26
units on a scale * year | 1.55 (2.02) | 0.80 (1.96) | 0.46 (1.93) | 0.89 (1.81) | 0.75 (1.82) | 1.30 (2.30)

2. Secondary Outcome: Slopes of 25 Foot Walk (25FW) Time
Description: slopes of measured times of 25FW during the 3-year 09-I-0197 trial (one year of pre-treatment baseline and two years of double-blind randomized treatment) and during one year extension phase of the 13-I-0088 trial. The slopes were measured separately for placebo and active treatment arm as randomized in the the 09-I-0197 trial.
  Lower extremity disability was measured by an average of two trials of timed 25 foot walk assessed every 6 month.
  The maximum time assigned for a trial is 180s. Patients unable to complete the 25 foot trial within this time limit are coded as "179.9"
Time Frame: 3-years double-blind phase and 1-year extension phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: seconds per year
Groups:
- Placebo Arm of the 09-I-0197: placebo arm of the 09-I-0197 - one year pre-treatment baseline plus two years of placebo during the double-blind phase of 09-I-0197
- Extension Phase (Placebo Arm): One-year open label extension phase of the 09-I-0917 placebo arm
- Active Treatment Arm of the 09-I-0197: active treatment arm of the 09-I-0197 - one year pre-treatment baseline plus two years of Idebenone treatment during the double-blind phase of 09-I-0197
- Extension Phase (Active Treatment Arm): One-year open label extension phase of the 09-I-0917 active treatment arm
Arm/Group | Placebo Arm of the 09-I-0197 | Extension Phase (Placebo Arm) | Active Treatment Arm of the 09-I-0197 | Extension Phase (Active Treatment Arm)
Number analyzed (Participants) | 30 | 22 | 31 | 26
seconds per year | 0.04322 (0.009617) | -0.00531 (0.01599) | 0.04031 (0.0106) | 0.03401 (0.01286)

3. Secondary Outcome: Slopes of 9 Hole Peg Test (9HPT) Time
Description: Slopes of measured times of 9HPT during the 3-year 09-I-0197 trial (one year of pre-treatment baseline and two years of double-blind randomized treatment) and during one year extension phase of the 13-I-0088 trial. The slopes were measured separately for placebo and active treatment arm as randomized in the the 09-I-0197 trial.
  Upper extremity/fine motor movements disability was measured as an average of left and right hand time, with each hand assessed as an average of two trials with upper limit of 5 (300s) per trial. Patients unable to complete the task within this time are coded as "777" The outcome was assessed every 6 months.
Time Frame: 3-years double-blind phase and 1-year extension phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: seconds per year
Arm/Group | Placebo Arm of the 09-I-0197 | Extension Phase (Placebo Arm) | Active Treatment Arm of the 09-I-0197 | Extension Phase (Active Treatment Arm)
Number analyzed (Participants) | 30 | 22 | 31 | 26
seconds per year | 0.000665 (0.000491) | 0.000947 (0.001189) | 0.000718 (0.000462) | 0.001086 (0.000614)

4. Secondary Outcome: Slopes of Expanded Disability Status Scale (EDSS) Score
Description: Slopes of measured EDSS scores during the 3-year 09-I-0197 trial (one year of pre-treatment baseline and two years of double-blind randomized treatment) and during one year extension phase of the 13-I-0088 trial. The slopes were measured separately for placebo and active treatment arm as randomized in the the 09-I-0197 trial.
  EDSS scale combines various elements of neurological exam. EDSS is a discrete scale ranging from 0 to 10 with 0.5 point increments. EDSS of 0 means no neurological disability, while EDSS of 10 marks death due to Multiple Sclerosis (MS). EDSS was assessed every 6 months.
Time Frame: 3-years double-blind phase and 1-year extension phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale per year
Arm/Group | Placebo Arm of the 09-I-0197 | Extension Phase (Placebo Arm) | Active Treatment Arm of the 09-I-0197 | Extension Phase (Active Treatment Arm)
Number analyzed (Participants) | 30 | 22 | 31 | 26
score on a scale per year | 0.1447 (0.05778) | 0.1435 (0.07625) | 0.1107 (0.03651) | 0.1584 (0.09479)

5. Secondary Outcome: Change in Slopes of Scripps Neurological Rating Scale (SNRS) Score
Description: Slopes of measured SNRS scores during the 3-year 09-I-0197 trial (one year of pre-treatment baseline and two years of double-blind randomized treatment) and during one year extension phase of the 13-I-0088 trial. The slopes were measured separately for placebo and active treatment arm as randomized in the the 09-I-0197 trial.
  SNRS scale combines various elements of a neurological exam into a single number. The scale ranges from 100 to 0, where 100 marks no disability and 0 marks maximum disability.
  SNRS was assessed every 6 months.
Time Frame: 3-years double-blind phase and 1-year extension phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale per year
Arm/Group | Placebo Arm of the 09-I-0197 | Extension Phase (Placebo Arm) | Active Treatment Arm of the 09-I-0197 | Extension Phase (Active Treatment Arm)
Number analyzed (Participants) | 30 | 22 | 31 | 26
score on a scale per year | -1.8838 (0.4829) | -2.1655 (1.0735) | -2.009 (0.3789) | -2.7263 (1.0073)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events are collected on 61 patients enrolled in the 1-year open-label phase
Groups:
- Active Treatment in 09-I-0197: Idebenone (150mg tablets) administered orally as five tablets, three times per day with food.
  Two years of Idebenone treatment during the 09-I-0197 double-blind phase
- Placebo in 09-I-0197: Idebenone (150mg tablets) administered orally as five tablets, three times per day with food.
  Two years of placebo during the 09-I-0197 double-blind phase
Arm/Group | Active Treatment in 09-I-0197 | Placebo in 09-I-0197
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/31 | 4/30
Other Adverse Events (participants affected / at risk) | 10/31 | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment in 09-I-0197 (N=31) | Placebo in 09-I-0197 (N=30)
Elevated liver enzynes (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
decreased ejection fraction (Cardiac disorders) | 1 (1) | 0 (0)
stomach cancer (Gastrointestinal disorders) | 0 (0) | 1 (1)
severe constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0)
ruptured apendix (Infections and infestations) | 0 (0) | 1 (1)
broken ribs (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
broken femur (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
chest tightness (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment in 09-I-0197 (N=31) | Placebo in 09-I-0197 (N=30)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
benign thyroid nodule (Endocrine disorders) | 0 (0) | 1 (1)
cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (2) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (2) | 6 (7)
fractured bone (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
hair loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
increased mobility problems (General disorders) | 0 (0) | 1 (1)
injured meniscus (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
penumonia (Infections and infestations) | 1 (1) | 0 (0)
radiculopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
retinal detachment (Eye disorders) | 0 (0) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
transient graying of vision (Eye disorders) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT01854359/Prot_SAP_000.pdf